CLINICAL TRIAL: NCT04101006
Title: Cerebrovascular Autoregulation During Major Non-cardiac Surgery and Risk for Postoperative Cognitive Dysfunction in Elderly Patients
Brief Title: Perioperative Changes of Cerebrovascular Autoregulation and Association With Cognitive Function
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties, high postoperative drop-out rate
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV4771
Record Dates: First submitted 2019-07-24; First posted 2019-09-24 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Function Abnormal; Anesthesia; Surgery
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral blood flow is tightly regulated to ensure constant cerebral perfusion independently from systemic blood pressure fluctuations. This mechanism is termed cerebrovascular autoregulation and preserves adequate cerebral perfusion in a range between 50 and 150 mmHg of cerebral perfusion pressure. Upper and lower autoregulatory limits may vary individually. Beyond the autoregulatory range the protective autoregulatory response is lost, facilitating cerebral ischemia or hyperemia.

The cerebrovascular response may be altered during general anesthesia, through direct effects of anesthetic agents on the vascular tone, changes of arterial partial pressure of carbon dioxide or the administration of vasoactive substances. The association of perioperative impairment of cerebral autoregulation and postoperative cognitive function has been discussed controversially.

DETAILED DESCRIPTION:
* continuous monitoring of cerebrovascular autoregulation using the correlation method
* based on near-infrared spectroscopy and invasive blood pressure measurement an index (COx) will be calculated
* autoregulation monitoring from anesthesia induction until emergence from anesthesia
* assessment of preoperative cognitive function during preanesthesia evaluation or on the day before surgery
* assessment of postoperative cognitive function between day 3 and 14 following surgery
* evaluation of subjective cognitive complaints or attention deficits 3 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* elective major non-cardiac/non-vascular surgery
* anticipated surgical duration >120 minutes
* age >= 60 years
* indication for invasive blood pressure measurement
* native German speaker

Exclusion Criteria:

* history of cerebrovascular disease
* preexisting cognitive impairment
* history or presence of neurological disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: screening of patients scheduled for preanesthesia evaluation prior to major non-cardiac/non-vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Postoperative change of cognitive function from baseline | preoperative psychometric evaluation on the day before surgery, postoperative psychometric evaluation between day 3 and 14 after surgery
  change of cognitive function following surgery compared with preoperative cognitive performance, defined as: z-score <-1.96/>1.96 in two or more neuropsychological tests (California Verbal Learning Test for verbal learning, Grooved Pegboard Test for visual motoric coordination, Digit Span forward task for attention and memory, Trail-Making-Test A and B for executive function) and/or a combined z-score >1.96

SECONDARY OUTCOMES:
cognitive failures three months following surgery | three months after elective surgery
  Self-assessment of cognitive failures using a validated questionnaire (Cognitive Failures Questionnaire). The questionnaire evaluates self-reported failures in perception, memory, and motor function. The questionnaire contains 25 items on a 5-point Likert scale. Total sum score from 0 (minimum) to 100 (maximum).

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fischer, MD, PhD, Principal Investigator — Department of Anesthesiology, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Kahl U, Rademacher C, Harler U, Juilfs N, Pinnschmidt HO, Beck S, Dohrmann T, Zollner C, Fischer M. Intraoperative impaired cerebrovascular autoregulation and delayed neurocognitive recovery after major oncologic surgery: a secondary analysis of pooled data. J Clin Monit Comput. 2022 Jun;36(3):765-773. doi: 10.1007/s10877-021-00706-z. Epub 2021 Apr 15. PMID 33860406